CLINICAL TRIAL: NCT05729282
Title: Role of Hyperinsulinemia in Non-Alcoholic Fatty Liver Disease (NAFLD) Pathogenesis: Diazoxide Pilot & Feasibility Study
Brief Title: Glycemic Effect of Diazoxide in NAFLD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of California, Berkeley (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AAAU2570; K12DK133995 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hyperinsulinemia; Insulin Resistance; Non-Alcoholic Fatty Liver Disease; Prediabetic State
Keywords: Insulin resistance; Hyperinsulinemia; Non-Alcoholic Fatty Liver Disease; Triglycerides
MeSH Terms: conditions — Hyperinsulinism; Insulin Resistance; Non-alcoholic Fatty Liver Disease; Prediabetic State | interventions — Diazoxide; Deuterium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both investigators and participants will be blinded to the assigned treatment group. Routine unblinding will occur to investigators only after all of a participant's samples have been submitted for laboratory analysis. It should be noted that investigators may get a sense of group allocation based on changes in blood glucose. However, due to interindividual variability in extent of insulin resistance and body mass index, it will not be possible to assuredly decode the randomization prior to unblinding. The blinding of the study Principal Investigator (PI) will be repealed only in the case of early withdrawal and/or medical emergency (e.g., severe hyperglycemia), which in most cases will result in study termination anyway. Participants will be notified of their group assignment once all relevant data are collected and analyzed if opted in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will ingest a placebo solution (27 doses over 14 days) formulated to approximate the taste of diazoxide oral suspension. Blinding will occur by completely covering single-dose oral syringes with labels.
  Interventions: Drug: Placebo; Device: FreeStyle Libre Pro; Drug: Deuterated water (2H2O/D2O)
- Diazoxide oral suspension, 1 mg per kg per dose (Experimental): Participants will ingest diazoxide oral suspension at 1 mg per kg body weight per dose (27 doses over 14 days). Blinding will occur by completely covering single-dose oral syringes with labels.
  Interventions: Drug: Diazoxide oral suspension, 1 mg per kg per dose; Device: FreeStyle Libre Pro; Drug: Deuterated water (2H2O/D2O)
- Diazoxide oral suspension, 2 mg per kg per dose (Experimental): Participants will ingest diazoxide oral suspension at 2 mg per kg body weight per dose (27 doses over 14 days). Blinding will occur by completely covering single-dose oral syringes with labels.
  Interventions: Drug: Diazoxide oral suspension, 2 mg per kg per dose; Device: FreeStyle Libre Pro; Drug: Deuterated water (2H2O/D2O)

INTERVENTIONS:
Drug: Diazoxide oral suspension, 1 mg per kg per dose — Diazoxide oral suspension provided in label-obscured single-use oral syringes at 1 mg per kg per dose (total of 27 doses over 14 days).
  Other Names: Proglycem
  Arms: Diazoxide oral suspension, 1 mg per kg per dose
Drug: Diazoxide oral suspension, 2 mg per kg per dose — Diazoxide oral suspension provided in label-obscured single-use oral syringes at 2 mg per kg per dose (total of 27 doses over 14 days).
  Other Names: Proglycem
  Arms: Diazoxide oral suspension, 2 mg per kg per dose
Drug: Placebo — Flavor-approximate placebo consisting of peppermint extract in diet tonic water, thickened with xanthan gum, provided in label-obscured single-use oral syringes at 2 mg per kg per dose (total of 27 doses over 14 days).
  Other Names: Placebo solution
  Arms: Placebo
Device: FreeStyle Libre Pro — All participants will wear a FreeStyle Libre Pro continuous glucose monitor (CGM) to track glycemic trends in response to study treatments. Investigators and participants will be blinded to CGM readings until after each participant has completed the trial.
Drug: Deuterated water (2H2O/D2O) — All participants will consume 32 aliquots of deuterated water (2H2O/D2O) 50 mL over 14 days to assess hepatic de novo lipogenesis. Tracer enrichment will be determined in blood and saliva.
  Other Names: Heavy water

SUMMARY:
The goal of this clinical trial is to compare a two-week course of diazoxide (at two different doses) and placebo in people with overweight/obesity and insulin resistance (IR) with, or at high risk for, non-alcoholic fatty liver disease (NAFLD). The main questions it aims to answer are how mitigation of compensatory hyperinsulinemia with diazoxide affects parameters of glucose and lipid metabolism (how people with IR and NAFLD respond to lowering high insulin levels so that the investigators can see what happens to how the liver handles fat and sugar).

Participants will:

* Take 27 doses of diazoxide (at 1 mg per kg of body weight per dose [mpk] or 2 mpk) or of placebo, over 14 days
* Take 32 doses of heavy (deuterated) water (50 mL each) over 14 days
* Have blood drawn and saliva collected after an overnight fast on four mornings over the two-week study period
* Consume their total calculated daily caloric needs as divided into three meals per day
* Wear a continuous glucose monitor for the two-week study period

Researchers will compare fasting blood tests at intervals during the study period in participants randomized (like the flip of a coin) to diazoxide 1 mpk, diazoxide 2 mpk, or placebo, to see how the drug treatment affects plasma glucose, serum insulin, and serum lipid parameters (triglycerides, free fatty acids, and apolipoprotein B). They will also consume heavy (deuterated) water to assess de novo lipogenesis (building of new fatty acids by the liver).

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is an under-appreciated complication of lipid dysmetabolism in type 2 diabetes (T2DM). Although it appears that insulin resistance (IR) is a mechanism common to both, the pathophysiology of its connection to unhealthy fat accumulation in the liver remains unclear. The investigators propose that the hyperinsulinemia that accompanies IR drives the excess hepatic de novo lipogenesis (DNL) that characterizes IR-associated NAFLD (IR-NAFLD). As such, despite its potential impact on glucose tolerance, lowering insulin levels might attenuate the pro-steatotic drive in patients with IR. The investigators' long-term objective, therefore, is to blunt endogenous insulin secretion using the insulin anti-secretagogue diazoxide in order to assess the impact on DNL. However, in order to optimize diazoxide treatment conditions, the investigators must first perform a pilot & feasibility study.

This is a single-center, randomized, double blinded, placebo-controlled clinical trial to provide pilot and feasibility data on the use of diazoxide oral suspension to ameliorate hyperinsulinemia in participants with overweight/obesity and insulin resistance (prediabetic state or elevated Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) score, + fasting hyperinsulinemia) who are diagnosed with, or clinically judged to be at high risk of, NAFLD. Participants will be randomized to one of three parallel arms: placebo, diazoxide at 1 mg per kg of body weight (mpk) per dose, or diazoxide at 2 mpk per dose, for a total of 27 doses over 14 days. They will also consume heavy (deuterated) water for a total of 32 doses of 50 ml over 14 days to measure de novo lipogenesis, an exploratory endpoint. They will present for outpatient blood draws and saliva collections after an overnight fast at four time points during the study course. Additionally, participants will follow a weight-maintaining diet and wear a professional continuous glucose monitor (CGM) throughout.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-70 years (using highly effective contraception if of childbearing potential)
2. Body mass index of 27-50 kg/m2
3. Able to understand written and spoken English and/or Spanish
4. Able to have pre-randomization screening labs drawn and study protocol initiated within 30 days of informed consent
5. Diagnosed with, or clinically judged to be at high risk for, non-alcoholic fatty liver disease (NAFLD), also known as metabolic-associated fatty liver disease (MAFLD), by hepatologist or other qualified physician
6. Evidence of insulin resistance, represented by any or all of the following criteria:

   i. Meeting either of the American Diabetes Association's definitions for prediabetes or IFG on screening labs:
   1. Prediabetes: Hemoglobin A1c 5.7-6.4%
   2. IFG: plasma glucose of 100-125 mg dL-1 after ≥ 8-h fast

   and/or

   ii. Homeostasis Model of Insulin Resistance (HOMA-IR) score ≥ 2.73
7. Fasting hyperinsulinemia (fasting insulin level ≥ 13 µIU/mL) on screening labs
8. Written informed consent (in English or Spanish) and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

1. Unable to provide informed consent in English or Spanish
2. Concerns arising at screening visit (any of the following):

   i. Documented weight loss of ≥ 5.0% of baseline within the previous 6 months

   ii. Abnormal blood pressure (including on treatment, if prescribed) • Systolic blood pressure < 95 mm Hg or > 160 mm Hg, and/or

   • Diastolic blood pressure < 65 mm Hg or > 100 mm Hg

   iii. Abnormal resting heart rate < 60 bpm or ≥ 100 bpm

   • Sinus brady- or tachycardia that has been appropriately evaluated and considered benign by the recruit's personal physician may be permitted at PI's discretion

   iv. Abnormal screening electrocardiogram (or if on file, performed within previous 90 d):
   * Non-sinus rhythm
   * Significant corrected QT segment (QTc) prolongation (≥ 480 ms)
   * New or previously unknown ischaemic changes that persist on repeat EKG:

     •• ST segment elevations

     •• T-wave inversions

     v. Laboratory evidence of diabetes mellitus:
   * Hemoglobin A1c ≥ 6.5%, and/or
   * Fasting plasma glucose ≥ 126 mg/dL

   vi. Positive qualitative serum β-hCG (human chorionic gonadotropin, beta subunit; i.e., pregnancy test) in women of childbearing potential

   vii. Liver function abnormalities
   * Transaminases (AST or ALT) > 3.0 x the upper limit of normal, and/or
   * Total bilirubin > 1.25 x the upper limit of normal

   viii. Abnormal screening triglycerides > 500 mg/dL

   ix. Abnormal screening serum electrolytes (any of the following) • Sodium, potassium, chloride, or bicarbonate levels that are considered clinically significant according to the clinical judgment of the PI • Creatinine equating to estimated glomerular filtration rate < 60 mL/min/1.73 m2

   x. Uric acid level above the upper limit of normal

   xi. Glucose-6-phosphate dehydrogenase below the lower limit of normal
3. COVID-19 precautions

   i. Unwillingness to comply with masking requirements per hospital policy

   ii. Active, documented COVID-19 at any time after screening
4. Reproductive concerns

   i. Women of childbearing potential not using highly effective contraception, defined as:
   * Surgical sterilization (e.g., bilateral tubal occlusion, bilateral oophorectomy and/or salpingectomy, hysterectomy)
   * Combined oral contraceptive pills taken daily, including during the study
   * Intrauterine device (levonorgestrel-eluting or copper) active at the time of the study
   * Medroxyprogesterone acetate (Depo-Provera®) injection active at the time of the study
   * Etonogestrel implants (e.g., Implanon®, etc.) active at the time of the study
   * Etonogestrel/ethinyl estradiol vaginal rings (e.g., Nuvaring®, etc.) active at the time of the study
   * Norelgestromin/ethinyl estradiol transdermal system (e.g., Ortho-Evra®) active at the time of the study

   ii. Women currently pregnant (tested by serum and/or urine β-hCG)

   iii. Women currently breastfeeding
5. Concerns related to glucose metabolism

   i. History of having met any of the American Diabetes Association's definitions of diabetes mellitus (i.e., overt diabetes):
   * Hemoglobin A1c ≥ 6.5%, or rapid rise in documented HbA1c values causing clinical concern for evolving insulin deficiency
   * Plasma glucose ≥ 126 mg/dL after 8-h fast
   * Plasma glucose of ≥ 200 mg/dL at 2 h after ingestion of a 75-g glucose load
   * Random plasma glucose ≥ 200 mg/dL associated with typical hyperglycemic symptoms, diabetic ketoacidosis, or hyperglycemic-hyperosmolar state

   ii. History of gestational diabetes mellitus within the previous 5 years

   iii. Use of most antidiabetic medications within the 90 days prior to screening
   * Excluded: thiazolidinediones, sulfonylureas, meglitinides, dipeptidyl peptidase-4 (DPP4) inhibitors, glucagon-like peptide 1 (GLP-1) receptor agonists, sodium-glucose cotransporter 2 (SGLT2) inhibitors, amylin mimetics, acarbose, insulin
   * Metformin is acceptable provided that recruits meet all of the inclusion criteria at screening

   iv. Clinical concern for absolute insulin deficiency (e.g., type 1 diabetes, pancreatic disease)
6. Concerns related to lipid metabolism

   i. Known diagnoses of familial hypercholesterolemia, familial combined hyperlipidemia, or familial hyperchylomicronemia

   ii. Use of certain lipid-lowering drugs within the 90 days prior to screening:
   * Statins or PCSK9 inhibitors for secondary prevention or for treatment of familial hypercholesterolemia. Statins or PCSK9 inhibitors for primary prevention of ASCVD are acceptable.
   * Fibrates (e.g., fenofibrate, clofibrate, gemfibrozil)
   * High-dose niacin (>100 mg daily)
7. Known, documented history (i.e., not to be newly screened/tested for study purposes), at the time of screening, of any of the following medical conditions:

   i. Pancreatic pathology, including but not limited to:
   * Pancreatic neoplasia, unless appropriately evaluated and considered benign and not producing hormones
   * Chronic pancreatitis
   * Acute pancreatitis within the previous 5 years
   * Autoimmune pancreatitis
   * Surgical removal of any portion of the pancreas

   ii. Cardiovascular disease (N.B. uncomplicated hypertension is not exclusionary)
   * Atherosclerotic cardiovascular disease
   * Stable or unstable angina
   * Myocardial infarction
   * Ischaemic or hemorrhagic stroke, or transient ischaemic attack
   * Peripheral arterial disease (claudication)
   * Use of dual antiplatelet therapy (aspirin + P2Y12 inhibitor)
   * History of percutaneous coronary intervention
   * Heart rhythm abnormalities
   * Congestive heart failure of any New York Heart Association class
   * Symptomatic valvular heart disease (e.g., aortic stenosis)
   * Pulmonary hypertension

   iii. Chronic kidney disease, Stage 3 or higher (estimated glomerular filtration rate < 60 mL/min/1.73 m2), of any cause

   iv. Chronic liver disease other than uncomplicated NAFLD, including but not limited to:
   * Advanced liver fibrosis, as determined by non-invasive testing
   * Cirrhosis of any etiology
   * Autoimmune hepatitis or other rheumatologic disorder affecting the liver
   * Biliopathy (e.g., progressive sclerosing cholangitis, primary biliary cholangitis)
   * Chronic liver infection (e.g., viral hepatitis, parasitic infestation)
   * Hepatocellular carcinoma
   * Infiltrative disorders (e.g., sarcoidosis, hemochromatosis, Wilson disease)

     v. Gout

   vi. Chronic viral illness (N.B. diagnosis based only on medical history; the investigators will not test for any of these viruses at any point in this study)
   * Hepatitis B virus (HBV), unless previously successfully eradicated with antiviral drugs that have been discontinued for at least 90 days prior to screening
   * Hepatitis C virus (HCV) infection, unless previously successfully eradicated with antiviral drugs that have been discontinued for at least 90 d prior to screening
   * Human immunodeficiency virus (HIV) infection

   vii. Malabsorptive conditions
   * Active inflammatory bowel disease (quiescent and off medication is acceptable)
   * Celiac disease (in remission on gluten-free diet is acceptable)
   * Surgical removal of a significant length of intestine

   viii. Active seizure disorder (including controlled with antiepileptic drugs)

   ix. Psychiatric diseases that:
   * Are or have been decompensated within 1 year of screening, and/or
   * Require use of anti-dopaminergic antipsychotic drugs associated with significant weight gain/metabolic dysfunction (e.g., clozapine, olanzapine), monoamine oxidase inhibitors, tricyclic antidepressants, or lithium

     x. Glucose-6-phosphate dehydrogenase (G6PD) deficiency
   * Due to presence of quinine in tonic water placebo

   xi. Other endocrinopathies:
   * Cushing syndrome (okay if considered in remission after treatment, provided that no exogenous corticosteroids are required)
   * Adrenal insufficiency
   * Primary aldosteronism

   xii. Venous thromboembolic disease (deep vein thrombosis or pulmonary embolism) or any required use of therapeutic anticoagulation

   xiii. Active malignancy, or hormonally active benign neoplasm, except allowances for:
   * Non-melanoma skin cancer
   * Differentiated thyroid cancer (AJCC Stage I only)
8. Clinical concern for increased risk of volume overload or hypotension (systolic blood pressure <95 and/or diastolic blood pressure <65 mm Hg), including due to medications and/or heart/liver/kidney problems, as listed above
9. Use of certain medications currently or within 90 d prior to screening:

   i. Prescribed medications used for any of the indications in the preceding list of excluded conditions, or their use within 90 d prior to screening, except allowances for:
   * Statins for primary prevention of cardiovascular disease
   * Use of drugs prescribed for indications other than the exclusionary diagnoses/purposes listed above (e.g., non-hydantoin antiepileptic drugs used for non-seizure indications, angiotensin converting enzyme inhibitors (ACEi)/angiotensin receptor blockers (ARB) used for uncomplicated hypertension rather than for congestive heart failure, etc.) •• Note, as above, that antidiabetic drugs for any indication (except metformin) within 90 d of screening are excluded

   ii. Vasodilating drugs for any indication: hydralazine, nitrates, phosphodiesterase-5 inhibitors (e.g., sildenafil, tadalafil), minoxidil (oral)

   iii. Phenytoin or fosphenytoin for any indication

   iv. Oral or parenteral corticosteroids (at greater than prednisone 5 mg daily, or equivalent) for more than 3 days within the previous 90 days; topical and inhaled formulations are permitted

   v. Fludrocortisone

   vi. Opioids
10. History of certain weight-loss (bariatric) surgeries, including:

    i. Roux-en-Y gastric bypass

    ii. Biliopancreatic diversion

    iii. Restrictive procedures (lap band, sleeve gastrectomy) performed within past 6 months
11. Clinical concern for alcohol overuse, including based on chart review and/or by participant's report of consuming more than 14 standard drinks per week for males or more than 7 standard drinks per week for females
12. Positive urine drug screen, except for:

    * Lawfully prescribed medication
    * Marijuana/THC positivity is okay, provided that the participant agrees not to use it during the same period that they will abstain from alcohol
13. History of severe infection or ongoing febrile illness within 30 days of screening
14. Any other disease or condition or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.
15. Known allergy/hypersensitivity to any component of the medicinal product formulations (including sulfa drugs), other biologics, IV infusion equipment, plastics, adhesive or silicone, history of infusion site reactions with IV administration of other medicines, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
16. Concurrent enrollment in another clinical study of any investigational drug therapy or use of any biologicals within 6 months prior to screening or within 5 half-lives of an investigational agent or biologic, whichever is longer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose (absolute values) | Up to Study Day 15
  Measurement of fasting plasma glucose levels during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: mg/dL).
Fasting plasma glucose (relative/change) | Up to Study Day 15
  Measurement of fasting plasma glucose during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: fold difference and/or Δmg/dL versus other groups).
Fasting plasma/serum insulin (absolute values) | Up to Study Day 15
  Measurement of fasting endogenous insulin levels during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: micro-international units [µIU] per mL).
Fasting plasma/serum insulin (relative change) | Up to Study Day 15
  Measurement of fasting endogenous insulin levels during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: fold difference and/or ΔµIU/mL versus other groups).

SECONDARY OUTCOMES:
Fasting serum or plasma triglycerides (TG) (absolute values) | Up to Study Day 15
  Measurement of fasting circulating TG during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: mg/dL).
Fasting serum/plasma triglycerides (TG) (relative/change) | Up to Study Day 15
  Measurement of fasting serum TG during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: fold difference and/or Δmg/dL versus other groups).
Fasting serum or plasma free fatty acids (FFA) (absolute values) | Up to Study Day 15
  Measurement of fasting serum FFA (units: mmol/L) during treatment with diazoxide 1 mpk vs 2 mpk vs placebo
Fasting serum or plasma free fatty acids (FFA) (relative/change) | Up to Study Day 15
  Measurement of fasting serum FFA during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: fold difference and/or Δmmol/L versus other groups)
Fasting serum/plasma apolipoprotein B (ApoB) (absolute values) | Up to Study Day 15
  Measurement of fasting serum/plasma ApoB during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: mg/dL)
Fasting serum/plasma apolipoprotein B (ApoB) (relative/change) | Up to Study Day 15
  Measurement of fasting serum/plasma ApoB during treatment with diazoxide 1 mpk vs 2 mpk vs placebo (units: mg/dL)
Continuous glucose monitoring (CGM) profile | Up to Study Day 15
  Measurement of interstitial glucose profiles during treatment with diazoxide 1 mpk vs 2 mpk vs placebo over the 2-week study course

OTHER OUTCOMES:
Hepatic de novo lipogenesis (absolute values) | Up to Study Day 15
  Percent incorporation of newly synthesized fatty acids into serum or VLDL TG (units: %)
Hepatic de novo lipogenesis (relative/change) | Up to Study Day 15
  Percent incorporation of newly synthesized fatty acids into serum or VLDL TG (units: fold difference and/or ∆% versus other groups)
Deuterium tracer enrichment in body water (measured in blood) | Up to Study Day 15
  Enrichment of total body water with deuterated water (2H2O/D2O) (units: %)
Deuterium tracer enrichment in body water (measured in saliva) | Up to Study Day 15
  Enrichment of total body water with deuterated water (2H2O/D2O) (units: %)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Blood samples will be banked in the Insulin Resistance Biobank and will be made available to other researchers for legitimate research purposes upon request. Associated data will be shared along with specimens in the smallest possible quantity and on a need-to-know basis. No Protected Health Information (PHI) will ever be disclosed to other researchers. All requests will be reviewed by the PI for scientific merit and samples/data will be transferred only upon completion of an Institutional Review Board (IRB)-approved Material Transfer Agreement (MTA) and/or Data Use Agreement (DUA), as appropriate.
Supporting Information: Study Protocol
Time Frame: Indefinitely following study completion.